CLINICAL TRIAL: NCT04491383
Title: Tocotrienols in Parkinson's Disease (PD): A Pilot, Randomised, Placebo-controlled Trial
Brief Title: Tocotrienols in Parkinson's Disease (PD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T3-PD-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Neuro-Degenerative Disease; Parkinson Disease
Keywords: Parkinson Disease; Vitamin E; Neurodegenerative Disease; Neurology
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: Experimental (Tocovid Suprabio (HOV-12020)) vs Control (Placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocovid Suprabio (HOV-12020) (Experimental): 200mg, twice 1 day, 12 months
  Interventions: Drug: Tocovid Suprabio (HOV-12020)
- Placebo (Placebo Comparator): 200mg, twice 1 day, 12 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tocovid Suprabio (HOV-12020) — Dietary supplement: Tocotrienol (HOV-12020) Palm oil-derived vitamin E, tocotrienol
  Arms: Tocovid Suprabio (HOV-12020)
Other: Placebo — Dietary supplement: Placebo. Placebo.
  Arms: Placebo

SUMMARY:
A study using Parkinson's disease animal model, transgenic fruit flies, demonstrated the potential of using tocotrienols (HOV-12020) as a therapeutic agent for delaying Parkinsonian motor dysfunctions. The proposed study aims to enrol 100 PD patients in a randomized placebo-controlled trial to investigate the effects of tocotrienols (HOV-12020) in motor and non-motor outcomes. Patients will be given oral tocotrienols (400mg/day) or placebo for 104 weeks. They will be assessed using the standard assessments scales in PD at baseline, Week 52 and Week 104. Neuropsychological evaluation will also be completed at these intervals to monitor progression of cognitive impairment (if any). Additional PD staging using MDSUPDRS (Part III), Hoehn & Yahr (H&Y) will be conducted at Week 26 and week 78. Blood samples will be collected to evaluate PD biomarkers and for safety monitoring (liver function, renal function and hematology).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 40 - 90 years (inclusive).
* Able to provide written informed consent and able to comply with study protocol.
* Idiopathic PD of more than 1 years duration from diagnosis. The diagnosis must be confirmed by presence of bradykinesia and at least 1 other cardinal sign (resting tremor, rigidity), without any other known or suspected cause of parkinsonism.
* Hoehn & Yahr => 2 with treatment.
* Patients on PD medication(s) e.g. levodopa, dopamine agonists, amantadine and/or Monoamine oxidase (MAO)-B inhibitors, must be on stable dose, for at least 30 days prior to screening. Medication and dose adjustments are allowed but must be documented.
* Patients on anti-depressant or anxiolytic medication must be on stable dose for at least 90 days prior to screening.
* The patient is willing to abstain from Vitamin E supplements (tocopherols and tocotrienols) and other dietary supplements which contain Vitamin E (tocopherols and tocotrienols) up to 14 days before baseline visit, and throughout the clinical study, unless prescribed by their physician for medical reasons.

Exclusion Criteria:

* Any other neurodegenerative disorder, such as Alzheimer's disease, Huntington's disease, or Creutzfeldt - Jakob disease.
* Current, clinically-significant hematological, cardiac, pulmonary, metabolic, neurologic or psychiatric disorders, uncontrolled seizures, untreated hypertension, disorders increasing risk of bleeding (Hemophilia), or any other significant active medical condition which, in the Investigator's opinion, would impact participation in this study.
* History of psychotic symptoms requiring treatment with a neuroleptic medication within the past 12 months.
* History of surgical or invasive intervention for PD (pallidotomy, thalamotomy, deep brain stimulation, etc.)
* Medical history indicating drug-induced parkinsonism (e.g., metoclopramide, flunarizine), metabolic identified neurogenetic disorders (e.g., Wilson's disease), encephalitis, or other atypical Parkinsonian syndromes (e.g., progressive supranuclear palsy, multiple system atrophy).
* History of myocardial infarction within 3 months prior to Screening, or current active angina pectoris, or symptomatic heart failure.
* Known liver disease or liver enzymes (AST, ALT) more than 5 times upper limit normal within 1 month of screening and enrolment.
* eGFR <60 within 1 month of screening and enrolment.
* Current participation in another investigational interventional study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline to Week 104 in Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Score | 104 weeks
  Score range is 0 to 199, with severity increasing with higher scores.

SECONDARY OUTCOMES:
Mean change from baseline to week 104 in disease severity | 104 weeks
Mean change from baseline to week 104 in individual cognitive domain z scores on comprehensive neuropsychological testing mean score change from baseline to week 104 in the MDS-UPDRS score for total score | 104 weeks
  Severity of disease increases with higher score.
Mean change from Baseline to Week 104 in quality of life, as measured by the Parkinson's Disease Questionnaire (PDQ-39) | 104 weeks
  Score range is 0 to 100. A lower score will indicate a better quality of life.
Difference proportion of patients with change from Baseline to Week 104, above or equal to the minimal clinically important difference (MCID) of the motor score, as measured by Part II and III subscales of MDS-UPDRS. | 104 weeks
  Severity of disease increases with higher score.
Mean change in levels of blood-based biomarkers (including total antioxidant status TAS, oxidative stress biomarkers and αsynuclein). | 104 weeks
Between treatment difference of type and incidence of Adverse Events (AEs) and Serious AEs (SAEs) | 104 weeks
Mean score change from Baseline to Week 104 in the MDS-UPDRS Part II scale | 104 weeks
  Severity of disease increases with higher score.
Mean score change from Baseline to Week 104 in the Schwab and England Activities of Daily Living (SE-ADL) scale. | 104 weeks
  The scale uses percentages to assess the difficulties completing daily activities/chores, from 0% to 100%. A higher percentage will indicate a better outcome (i.e. more independence for an individual).

CONTACTS AND LOCATIONS:
Overall Officials: Eng King Tan, Principal Investigator — National Neuroscience Institute Singapore; Adeline Su-Lyn Ng, Principal Investigator — National Neuroscience Institute Singapore
Locations (2):
- Singapore (2):
  - National Neuroscience Institute, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Gandhi S, Wood NW. Molecular pathogenesis of Parkinson's disease. Hum Mol Genet. 2005 Sep 15;14(18):2749-55. doi: 10.1093/hmg/ddi308. Epub 2005 Aug 26. PMID 16126732
- [Background] Khanna S, Rink C, Ghoorkhanian R, Gnyawali S, Heigel M, Wijesinghe DS, Chalfant CE, Chan YC, Banerjee J, Huang Y, Roy S, Sen CK. Loss of miR-29b following acute ischemic stroke contributes to neural cell death and infarct size. J Cereb Blood Flow Metab. 2013 Aug;33(8):1197-206. doi: 10.1038/jcbfm.2013.68. Epub 2013 May 1. PMID 23632968
- [Background] Rink C, Christoforidis G, Khanna S, Peterson L, Patel Y, Khanna S, Abduljalil A, Irfanoglu O, Machiraju R, Bergdall VK, Sen CK. Tocotrienol vitamin E protects against preclinical canine ischemic stroke by inducing arteriogenesis. J Cereb Blood Flow Metab. 2011 Nov;31(11):2218-30. doi: 10.1038/jcbfm.2011.85. Epub 2011 Jun 15. PMID 21673716
- [Background] Silbert LC, Howieson DB, Dodge H, Kaye JA. Cognitive impairment risk: white matter hyperintensity progression matters. Neurology. 2009 Jul 14;73(2):120-5. doi: 10.1212/WNL.0b013e3181ad53fd. PMID 19597134
- [Background] Srikanth VK, Quinn SJ, Donnan GA, Saling MM, Thrift AG. Long-term cognitive transitions, rates of cognitive change, and predictors of incident dementia in a population-based first-ever stroke cohort. Stroke. 2006 Oct;37(10):2479-83. doi: 10.1161/01.STR.0000239666.46828.d7. Epub 2006 Aug 31. PMID 16946165
- [Background] Sen CK, Rink C, Khanna S. Palm oil-derived natural vitamin E alpha-tocotrienol in brain health and disease. J Am Coll Nutr. 2010 Jun;29(3 Suppl):314S-323S. doi: 10.1080/07315724.2010.10719846. PMID 20823491
- [Background] Kuhad A, Chopra K. Tocotrienol attenuates oxidative-nitrosative stress and inflammatory cascade in experimental model of diabetic neuropathy. Neuropharmacology. 2009 Sep;57(4):456-62. doi: 10.1016/j.neuropharm.2009.06.013. Epub 2009 Jun 23. PMID 19555701
- [Background] Khanna S, Roy S, Slivka A, Craft TK, Chaki S, Rink C, Notestine MA, DeVries AC, Parinandi NL, Sen CK. Neuroprotective properties of the natural vitamin E alpha-tocotrienol. Stroke. 2005 Oct;36(10):2258-64. doi: 10.1161/01.STR.0000181082.70763.22. Epub 2005 Sep 15. PMID 16166580
- [Background] Khanna S, Roy S, Ryu H, Bahadduri P, Swaan PW, Ratan RR, Sen CK. Molecular basis of vitamin E action: tocotrienol modulates 12-lipoxygenase, a key mediator of glutamate-induced neurodegeneration. J Biol Chem. 2003 Oct 31;278(44):43508-15. doi: 10.1074/jbc.M307075200. Epub 2003 Aug 13. PMID 12917400
- [Background] Sen CK, Khanna S, Roy S, Packer L. Molecular basis of vitamin E action. Tocotrienol potently inhibits glutamate-induced pp60(c-Src) kinase activation and death of HT4 neuronal cells. J Biol Chem. 2000 Apr 28;275(17):13049-55. doi: 10.1074/jbc.275.17.13049. PMID 10777609
- [Background] Khanna S, Parinandi NL, Kotha SR, Roy S, Rink C, Bibus D, Sen CK. Nanomolar vitamin E alpha-tocotrienol inhibits glutamate-induced activation of phospholipase A2 and causes neuroprotection. J Neurochem. 2010 Mar;112(5):1249-60. doi: 10.1111/j.1471-4159.2009.06550.x. Epub 2009 Dec 17. PMID 20028458
- [Background] Aggarwal BB, Sundaram C, Prasad S, Kannappan R. Tocotrienols, the vitamin E of the 21st century: its potential against cancer and other chronic diseases. Biochem Pharmacol. 2010 Dec 1;80(11):1613-31. doi: 10.1016/j.bcp.2010.07.043. Epub 2010 Aug 7. PMID 20696139
- [Background] Vitamin E in Neuroprotection Study (VENUS) Investigators; Hor CP, Fung WY, Ang HA, Lim SC, Kam LY, Sim SW, Lim LH, Choon WY, Wong JW, Ch'ng ASH, Beh KKM, Wee HC, Ong LM, Khan NAK, Sulaiman SAS, Shuaib IL, Bakar A, Yusof Y, Yusof YM, Abu Bakar F, Tang WS, Teh HL, Wahid NA, Saaidin S, Idris N, Yoon CK, Ong HN, Ganapathy JT, Loo CE, Samy MM, Zainal H, Dharan SCS, Ooi BY, Teoh PY, Tye YL, Yeoh CA, Low DW, Looi I, Yuen KH. Efficacy of Oral Mixed Tocotrienols in Diabetic Peripheral Neuropathy: A Randomized Clinical Trial. JAMA Neurol. 2018 Apr 1;75(4):444-452. doi: 10.1001/jamaneurol.2017.4609. PMID 29379943
- [Result] Farooqui T, Farooqui AA. Lipid-mediated oxidative stress and inflammation in the pathogenesis of Parkinson's disease. Parkinsons Dis. 2011 Feb 15;2011:247467. doi: 10.4061/2011/247467. PMID 21403820
- [Result] Gopalan Y, Shuaib IL, Magosso E, Ansari MA, Abu Bakar MR, Wong JW, Khan NA, Liong WC, Sundram K, Ng BH, Karuthan C, Yuen KH. Clinical investigation of the protective effects of palm vitamin E tocotrienols on brain white matter. Stroke. 2014 May;45(5):1422-8. doi: 10.1161/STROKEAHA.113.004449. Epub 2014 Apr 3. PMID 24699052